

#### A collaborative project between:

University of Alabama at Birmingham;
Weill Cornell Medical College of Cornell University;
University of Carolina at Chapel Hill;
East Carolina University;
North Carolina Area Health Education Centers;
Alabama Area Health Education Centers;
Health and Wellness Education Center of Livingston, AL;
West Central Alabama Community Health Improvement League of Camden,
AL;

ConnectionHealth, Birmingham, AL;
Open Water Coaching and Consulting, Cape Carteret, NC;
and 80 primary care practices,
peer coaches,
and practice facilitators living in the Black Belt region

Funded by NHLBI UH3 HL130691-05

### **Study Protocol**

Version November 1, 2021 NCT02866669 Unique Protocol ID: X160722009

# Southeastern Collaboration to Improve Blood Pressure Control in the US Black Belt – Addressing the Triple Threat

Statistical analysis plan: The main hypothesis test was at the individual patient level, adjusting for baseline covariates with imbalance across treatment arms and accounting for clustering using generalized estimating equations (GEE). Each intervention, alone or in combination, was compared to the enhanced usual care arm with p<0.05 serving as the threshold for statistical significance. To test for differences between trial arms we used the Benjamini-Hochburg approach to control the false-discovery rate at 0.05. The secondary outcome was change in systolic blood pressure levels, which was analyzed using linear regression adjusting for characteristics that were imbalanced across trial arms, state (AL vs. NC), and days from baseline to follow-up. All analyses accounted for clustering of patients within practices.

# Table 1. Adjusted Odds ratios (95% CI) for blood pressure control at 12 months, by trial arm compared to enhanced usual care

| Arm | 12 month OR (95% CI) |
|--------------|----------------------|
| PF vs. EUC | 0.97 (0.6, 1.58) |
| PC vs. EUC | 1.3 (0.83, 2.04) |
| PFPC vs. EUC | 1.02 (0.64, 1.64) |

Abbreviations: CI- confidence interval; EUC-enhanced usual care; PF-practice facilitation; PC-peer coaching; PFPC- practice facilitation and peer coaching.

a. Adjusts for baseline SBP, DBP, PHQ8, age, state, insurance, current smoking, health literacy.

## Table 2. Adjusted<sup>a</sup> Changes (95% CI) in systolic blood pressure at 12 months, by trial arm compared with enhanced usual care

| Arm | 12-month Diff. (95% CI) |
|--------------|-------------------------|
| PF vs. EUC | -0.08 (-4.07, 3.91) |
| PC vs. EUC | -2.34 (-6.06, 1.38) |
| PFPC vs. EUC | -2.06 (-5.94, 1.82) |

Abbreviations: CI- confidence interval; EUC-enhanced usual care; PF-practice facilitation; PC-peer coaching; PFPC- practice facilitation and peer coaching.

a. Adjusts for baseline SBP, DBP, PHQ8, age, state, insurance, current smoking, health literacy.

#### 44 Table 3. Adjusted differences (95% CI) for change in Physical Component Summary (PCS) score at 12 months

| Δ | | | |
|--------------|----------------|------------------------------------|------|
| Arm | n <sup>b</sup> | n <sup>b</sup> Coefficient (95%CI) | |
| EUC | 312 | ref | ref |
| PF vs. EUC | 236 | -1.59 (-2.96,-0.21) | 0.02 |
| PC vs. EUC | 309 | -0.15 (-1.43,1.13) | 0.82 |
| PFPC vs. EUC | 249 | -0.02 (-1.36,1.33) | 0.98 |

Abbreviations: CI- confidence interval; EUC-enhanced usual care; PF-practice facilitation; PC-peer coaching; PFPC- practice facilitation and peer coaching

- a. Adjusts for baseline PCS, SBP, DBP, PHQ8, age, state, insurance, current smoking, health literacy.
- b. N reflects complete case numbers in adjusted model; <1% of sample missing information on covariates.

Abbreviations: ppt-participant; CI-confidence interval; EUC-enhanced usual care; PF-practice facilitation; PC-

b. Total n reflects complete case numbers in fully adjusted model. <1% of sample missing information on co-

a. Adjusts for baseline MCS, SBP, DBP, age, state, insurance, PHQ-8, current smoking, and health literacy.

12 months

Coefficient (95%CI)

Ref

-0.30 (-2.09, 1.49)

0.54 (-1.11,2.20)

0.81 (-0.93, 2.55)

p-value

Ref

0.74

0.52

0.36

56

Arm

**EUC** 

PF vs. EUC

PC vs. EUC

PFPC vs. EUC

67

68

69

70

71

72

73 74

75

76

variates.

peer coaching; PFPC-practice facilitation and peer coaching.

Total n pptb

312

236

309

249

| Auss | 12 months | | |
|--------------|----------------|---------------------|---------|
| Arm | n <sup>b</sup> | Coefficient (95%CI) | p-value |
| EUC | 312 | ref | ref |
| PF vs. EUC | 238 | -0.10 (-0.60,0.39) | 0.68 |
| PC vs. EUC | 313 | -0.46 (-0.92,0.00) | 0.05 |
| PFPC vs. EUC | 249 | -0.22 (-0.70,0.26) | 0.36 |

Abbreviations: ppt-participant; Cl-confidence interval; EUC-enhanced usual care; PF-practice facilitation; PCpeer coaching; PFPC-practice facilitation and peer coaching.

- a. Adjusts for baseline PSS, baseline SBP, baseline DBP, age, state, insurance, PHQ-8, current smoking, health literacy
- b. Total n reflects complete case numbers in fully adjusted model. <1% of sample missing information on covariates

Table 6. Adjusted differences (95% CI) in change in patient assessment of chronic illness care (PACIC) at 12months

| Aum | 12 months | | |
|--------------|----------------|---------------------|---------|
| Arm | n <sup>b</sup> | Coefficient (95%CI) | p-value |
| EUC | 281 | ref | ref |
| PF vs. EUC | 221 | -0.00 (-0.21,0.20) | 0.97 |
| PC vs. EUC | 298 | 0.18 (-0.01,0.37) | 0.06 |
| PFPC vs. EUC | 230 | 0.24 (0.04,0.44) | 0.02 |

Abbreviations: ppt-participant; CI-confidence interval; EUC-enhanced usual care; PF-practice facilitation; PCpeer coaching; PFPC-practice facilitation and peer coaching.

a. Adjusts for PACIC, baseline SBP, baseline DBP, age, state, insurance, PHQ-8, current smoking, health literacy. b. Total n reflects complete case numbers in fully adjusted model. <1% of sample missing information on co-

77

78

Table 7. Adjusted odds ratios (95% CI) for ED visits at 12 months

| Λ | 12 months | | |
|--------------|---------------------|------------------|---------|
| Arm | Events/total n pptb | OR (95% CI) | p-value |
| EUC | 78/320 | ref | ref |
| PF vs. EUC | 57/243 | 0.91 (0.53,1.56) | 0.73 |
| PC vs. EUC | 65/317 | 0.72 (0.43,1.20) | 0.21 |
| PFPC vs. EUC | 55/260 | 0.77 (0.45,1.32) | 0.34 |

Abbreviations: ED-emergency department; ppt-participant; CI-confidence interval; EUC-enhanced usual care; PF-practice facilitation; PC-peer coaching; PFPC-practice facilitation and peer coaching; PHQ-8-patient health questionnaire depression scale.

- a. Adjusts for baseline ED (Y/N), baseline SBP, baseline DBP, age, state, insurance, PHQ-8, current smoking, health literacy.
- b. Total n reflects complete case numbers in fully adjusted model. <1% of sample missing information on covariates. c. Poor health literacy defined as having problems learning about conditions because can't understand written information a little to all of the time.

Table 8. Adjusted odds ratios (95% CI) for hospitalization at 12-months

| A 11110 | 12 months | | |
|--------------|---------------------|------------------|---------|
| Arm | Events/total n pptb | OR (95% CI) | p-value |
| EUC | 23/320 | ref | ref |
| PF vs. EUC | 35/243 | 2.19 (1.17,4.10) | 0.01 |
| PC vs. EUC | 31/317 | 1.37 (0.74,2.55) | 0.32 |
| PFPC vs. EUC | 30/260 | 1.78 (0.95,3.33) | 0.07 |

Abbreviations: ppt-participant; CI-confidence interval; EUC-enhanced usual care; PF-practice facilitation; PC-peer coaching; PFPC-practice facilitation and peer coaching; PHQ-8-patient health questionnaire depression scale.

- a. Adjusts for baseline hospitalization (Y/N), baseline SBP, baseline DBP, age, state, insurance, PHQ-8, current smoking, health literacy.
- b. Total n reflects complete case numbers in fully adjusted model. <1% of sample missing information on covariates.